CLINICAL TRIAL: NCT02337543
Title: NEO6860: A Phase I, Double-Blind, Placebo-Controlled, Single and Multiple Oral Dose, Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Study in Healthy Male and Female Subjects
Brief Title: NEO6860, a TRPV1 Antagonist, First in Human Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neomed Institute (Other)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEO6860-1301
Record Dates: First submitted 2015-01-09; First posted 2015-01-13 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2015-10

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active: NEO6860 (Experimental): NEO6860 suspension is the drug under evaluation
  Interventions: Drug: NEO6860
- placebo (Placebo Comparator): Placebo matching NEO6860 suspension formulation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NEO6860 — NEO6860 is an NCE acting as a TRPV1 antagonist
  Arms: Active: NEO6860
Drug: Placebo — Placebo
  Arms: placebo

SUMMARY:
This study is a double blind, placebo controlled, ascending single and multiple oral dose study conducted in two parts, aimed at determining the safety and tolerability of single and multiple oral doses of NEO6860 in healthy subjects.

Key secondary objectives are: assessment of the pharmacokinetic profile, effect of food and gender.

The analgesic effect of NEO6860 will be investigated using experimental capsaicin-evoked pain methods.

Part A will comprise an ascending single dose, with 6 dose levels. Part B will comprise an ascending multiple dose, with 2 dose levels.

DETAILED DESCRIPTION:
This study is a double blind, placebo controlled, ascending single and multiple oral dose study conducted in two parts, aimed at determining the safety and tolerability of single and multiple oral doses of NEO6860 in healthy subjects.

Key secondary objectives are: assessment of the pharmacokinetic profile, effect of food and gender.

The analgesic effect of NEO6860 will be investigated using experimental capsaicin-evoked pain methods. Measurement of capsaicin evoked pain, and secondary hyperalgesia will be performed at baseline and at estimated Tmax and 8 hours post dosing.

Part A will comprise an ascending single dose, sequential group study in male subjects, incorporating a two-period crossover group to investigate the effect of food and a single group of female subjects to investigate gender effect.

56 subjects will be studied in 7 groups (Groups A1 to A7), each group consisting of 8 subjects (6 subjects will receive NEO6860 and 2 will receive placebo). Six dose levels will be explored: 50, 100, 200, 400, 800 and 1 600mg.

Part B will comprise an ascending multiple dose, sequential group study. 16 subjects will be studied in 2 groups (Groups B1 to B2), each group consisting of 8 subjects (6 subjects will receive NEO6860 and 2 will receive placebo) receiving 5 days of therapy with a dose schedule to be determined during Part A.

ELIGIBILITY:
Inclusion Criteria:

Males and females Any ethnic origin Between 18 and 55 years of age Body mass index (BMI) between 18.0 and 32.0 kg/m2 inclusive Body weight between 50 kg and 100 kg inclusive Subjects must be in good health, as determined by Medical history, Physical examination, Vital sign assessment, 12-lead electrocardiogram (ECG), Clinical laboratory evaluations (congenital non-haemolytic hyperbilirubinaemia is acceptable) Subjects will have given their written informed consent to participate in the study and to abide by the study restrictions

Exclusion Criteria:

Male subjects who are not willing, or whose partners are not willing, to use appropriate contraception (such as a condom with spermicidal foam/gel/film/cream/suppository), or to refrain from donating sperm from the time of the first dose until 3 months after the final dosing occasion.

Subjects who have donated blood in the 3 months prior to screening, plasma in the 7 days prior to screening or platelets in the 6 weeks prior to screening Subjects who consume more than 28 units of alcohol per week if male or consume more than 21 units of alcohol per week if female

Subjects who have used any medication within 7 days of the first dose administration, unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise safety:

Subjects who have a clinically significant pulse rate, blood pressure or temperature that, in the opinion of the investigator, increases the risk of participating in the study, in accordance with the CRU reference ranges at screening and prior to first dose Subjects with a positive urine drug screen (confirmed by repeat) at screening or first admission, or a positive alcohol breath test result (confirmed by repeat) at screening or first admission Subjects who have an abnormality in the 12-lead ECG that, in the opinion of the investigator, increases the risk of participating in the study, in accordance with the CRU reference ranges at screening Subjects with, or with a history of, any clinically significant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychiatric, respiratory, metabolic, endocrine, haematological or other major disorders as determined by the Investigator ALT or AST >1.5 times ULN at screening and/or prior to first dose, confirmed by repeat testing Subjects considered non-acceptable responders to the intradermal capsaicin test at screening, defined as maximum VAS score of <3 or 10 Subjects who, in the opinion of the Investigator, should not participate in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of NEO6860 in healthy subjects | 10 days

SECONDARY OUTCOMES:
Pharmacokinetics of NEO6860 in healthy subjects | 10 days
Food effect on Pharmacokinetics of NEO6860 in healthy subjects | 10 days
Gender effect on Pharmacokinetics of NEO6860 in healthy subjects | 10 days
Pharmacodynamics effect (ID Capsaicin test) of NEO6860 in healthy subjects | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Dan A Chiche, MD, Study Director — Neomed Institute
Locations (1):
- Covance Cru, Leeds, United Kingdom

REFERENCES:
- [Derived] Brown W, Leff RL, Griffin A, Hossack S, Aubray R, Walker P, Chiche DA. Safety, Pharmacokinetics, and Pharmacodynamics Study in Healthy Subjects of Oral NEO6860, a Modality Selective Transient Receptor Potential Vanilloid Subtype 1 Antagonist. J Pain. 2017 Jun;18(6):726-738. doi: 10.1016/j.jpain.2017.01.009. Epub 2017 Feb 8. PMID 28188907